CLINICAL TRIAL: NCT00633568
Title: A Phase III Randomised Study Comparing Concomitant Radiochemotherapy With Cisplatin and Docetaxel as Induction Versus Consolidation Treatment in Patients With Locally Advanced Unresectable Non-small Cell Lung Cancer.
Brief Title: Randomised Study of Concomitant Radiochemotherapy in Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: European Lung Cancer Working Party (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ELCWP 01063
Record Dates: First submitted 2008-03-05; First posted 2008-03-12 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Non-small Cell Lung Carcinoma
Keywords: Non-small cell lung carcinoma; Concomitant radiochemotherapy; Cisplatin; Docetaxel; Radiotherapy; Chemotherapy; Unresectable stage III non-small cell lung carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): One course of chemotherapy with cisplatin and docetaxel followed by induction chemoradiotherapy followed by two courses of consolidation chemotherapy
  Interventions: Drug: Concomitant Radiochemotherapy - Radiotherapy 66 Gy, Cisplatin, and Docetaxel
- B (Experimental): Three courses of induction chemotherapy followed by consolidation chemoradiotherapy
  Interventions: Drug: Concomitant Chemoradiotherapy - Radiotherapy 66 Gy, Cisplatin, and Docetaxel

INTERVENTIONS:
Drug: Concomitant Radiochemotherapy - Radiotherapy 66 Gy, Cisplatin, and Docetaxel — Concurrent chemoradiotherapy: Radiotherapy 66 Gy in 2 Gy/fraction, 5 fractions/wk (6.5 weeks)with Cisplatin 20 mg/m²/week (6 times, beginning on day 1 of radiotherapy)and Docetaxel 20 mg/m²/week (6 times, beginning on day 1 of radiotherapy) Chemotherapy : Cisplatin 60 mg/m² and Docetaxel 75 mg/m² on day 1
  Arms: A
Drug: Concomitant Chemoradiotherapy - Radiotherapy 66 Gy, Cisplatin, and Docetaxel — Concurrent chemoradiotherapy: Radiotherapy 66 Gy in 2 Gy/fraction, 5 fractions/wk (6.5 weeks)with Cisplatin 20 mg/m²/week (6 times, beginning on day 1 of radiotherapy)and Docetaxel 20 mg/m²/week (6 times, beginning on day 1 of radiotherapy) Chemotherapy : Cisplatin 60 mg/m² and Docetaxel 75 mg/m² on day 1
  Arms: B

SUMMARY:
The purpose of the present trial is to assess if induction concurrent chemoradiotherapy followed by consolidation chemotherapy will improve survival in comparison with the same chemotherapy given as induction followed by consolidation concurrent chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of non-small cell carcinoma of the lung
* Initially unresectable non-metastatic stage III disease
* Availability for participating in the detailed follow-up of the protocol
* Presence of an evaluable or measurable lesion
* Written informed consent
* No functional or anatomical contraindication to chest irradiation

Exclusion Criteria:

* Prior treatment with chemotherapy, radiotherapy or surgery
* Performance status < 60 on the Karnofsky scale
* History of prior malignant tumour, except non-melanoma skin cancer or in situ carcinoma of the cervix or cured malignant tumour (more than 5 year disease-free interval)
* Neutrophils < 2,000/mm³
* Platelet cells < 100,000/mm3
* Serum bilirubin > 1.5 mg/100 ml
* Hepatic disease contra-indicating the administration of docetaxel and/or GOT or GPT ≥ 2.5x the normal value and/or alkaline phosphatase ≥ 5x the normal value
* Serum creatinine > 1.5 mg/100 ml and/or creatinine clearance < 60 ml/min
* Recent myocardial infarction (less than 3 months prior to date of diagnosis) or uncontrolled angina pectoris
* Congestive cardiac failure or cardiac arrhythmia requiring medical treatment
* Uncontrolled infectious disease
* Symptomatic polyneuropathy
* Auditive impairment contra-indicating cisplatin administration
* Serious medical or psychological factors which may prevent adherence to the treatment schedule
* Malignant pleural or pericardial effusion
* Homolateral supraclavicular lymph node excepting upper lobe lesion
* Heterolateral supraclavicular lymph node
* Known hypersensitivity to docetaxel or cisplatin
* Pregnancy or for pre-menopausal patient, incapacity to use adequate contraceptive method

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2007-01; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Survival | Survival will be dated from the day of randomisation until death or last follow up

SECONDARY OUTCOMES:
Response rate | At the end of the whole treatment
Toxicity | After each course of chemotherapy and at the end of treatment
Local control rate | After completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Berghmans, MD, Study Chair — European Lung Cancer Working Party
Locations (19):
- Belgium (11):
  - Department of Pneumology RHMS Hôpital de la Madeleine, Ath
  - Department of Pneumology Clinique Saint-Luc, Bouge
  - Department of Pneumology CHR St Joseph-Warquignies, Boussu
  - Department of Intensive Care Unit and Thoracic Oncology Institut Jules Bordet, Brussels
  - Department of Pneumology Hospital Ixelles-Molière, Brussels
  - Department of Pneumology CHU Charleroi, Charleroi
  - Department of Pneumology Hôpital Saint-Joseph, Gilly
  - Hôpital Ambroise Paré, Mons
  - Hôpital Vésale - Montigny-le-Tilleul, Montigny-le-Tilleul
  - Department of Pneumology Centre Hospitalier de Mouscron, Mouscron
  - CH Peltzer-La Tourelle, Verviers
- France (6):
  - Service de Pneumologie Centre Hospitalier de Douai, Douai
  - Service de Pneumologie Hôpital de Hayange, Hayange
  - Pneumology department of CHU Lille, Lille
  - Service de Pneumologie Centre Hospitalier Intercommunal le Raincy-Montfermeil, Montfermeil
  - Service de Pneumologie CHG Tourcoing, Tourcoing
  - Cabinet médical Saint-Michel, Valenciennes
- Medical Oncology St Savas Hospital, Athens, Greece
- Medical Oncology Hospital de Sagunto, Valencia, Spain

REFERENCES:
- See also: Click here for more information on the protocol — http://www.elcwp.org